CLINICAL TRIAL: NCT07059065
Title: A Post-market, Prospective, Controlled, Multicenter Clinical Study to Evaluate Radiographic Fusion of FIBERGRAFT™ Aeridyan Matrix Bone Graft Substitute in Subjects Who Undergo a Lumbar Posterolateral Fusion Surgery
Brief Title: FIBERGRAFT Aeridyan Posterolateral Fusion Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Synthes Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSS202303; DSS202303 (Other: DePuy Synthes Products, Inc.)
Record Dates: First submitted 2025-06-19; First posted 2025-07-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Degenerative Spine Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Confidentiality of subject data will be maintained by both the site and the sponsor in accordance with the local regulations. Data protection consent will be obtained from subjects as part of the informed consent process or within a separate HIPAA document if required by local procedures. The data submitted to the sponsor will be pseudonymized, and subjects will not be identified by name or other identifiable information such as date of birth (DOB). Each subject will be assigned a specific subject identification number beginning with the site number and a consecutive subject number. The collection, use, and disclosure of all personal data, including subject health and medical information, are to be maintained in compliance with applicable personal data protection and security laws and regulations that govern protected health information and their informed consent given by each clinical study subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Cohort A) (Experimental): Arm 1: 79 subjects (Cohort A) treated with FIBERGRAFT Aeridyan Matrix bone graft substitute in a 1 to 3 level instrumented lumbar posterolateral fusion including up to 2 consecutive levels of a posterior lumbar interbody fusion between L1-S1.
  Cohort A will have a score range of 6 - 14.5
  Interventions: Device: FIBERGRAFT™ Aeridyan Matrix Bone Graft Substitute
- Cohort B (Experimental): Arm 2: 79 subjects (Cohort B) treated with FIBERGRAFT Aeridyan Matrix bone graft substitute in a 1 to 3 level instrumented lumbar posterolateral fusion including up to 2 consecutive levels of a posterior lumbar interbody fusion between L1-S1.
  Cohort B will have a score range of 14.6 - 43.5
  Interventions: Device: FIBERGRAFT™ Aeridyan Matrix Bone Graft Substitute
- Controlled Cohort A (Active Comparator): Arm 3: 79 subjects (Cohort A) treated with Demineralized Bone Matrix in a 1 to 3 level instrumented lumbar posterolateral fusion including up to 2 consecutive levels of a posterior lumbar interbody fusion between L1-S1.
  Cohort A will have a score range of 6 - 14.5
  Interventions: Device: Demineralized Bone Matrix
- Controlled Cohort B (Active Comparator): Arm 4: 79 subjects (Cohort B) treated with Demineralized Bone Matrix in a 1 to 3 level instrumented lumbar posterolateral fusion including up to 2 consecutive levels of a posterior lumbar interbody fusion between L1-S1.
  Cohort B will have a score range of 14.6 - 43.5
  Interventions: Device: Demineralized Bone Matrix

INTERVENTIONS:
Device: FIBERGRAFT™ Aeridyan Matrix Bone Graft Substitute — FIBERGRAFT™ Aeridyan Matrix is a next generation synthetic bone graft that is resorbable, bioactive, and osteoconductive. FIBERGRAFT Aeridyan Matrix is composed of ultra-porous 45S5 bioactive glass granules, boron-based bioactive glass microspheres, and bovine type 1 collagen. The granules are made entirely of 45S5 bioactive glass fibers and feature a porous outer shell encasing an intricate nest of micro- and nano- fibers and microspheres. The nonporous microspheres are made entirely of boron-based bioactive glass and feature essential metallic ions such as zinc, copper, magnesium, and potassium. The highly biocompatible type 1 collagen5 serves as a carrier for the bioactive glass components.
  FIBERGRAFT Aeridyan Matrix is designed to have an adequate structural integrity for its application as a bone graft substitute material, while optimizing radiopacity and resorption.
  Arms: Cohort A); Cohort B
Device: Demineralized Bone Matrix — Demineralized Bone Matrix is to be used with bone marrow aspirate and mixed with autograft bone in accordance with approved indications per the IFU
  Arms: Controlled Cohort A; Controlled Cohort B

SUMMARY:
This is a post-market, prospective, controlled, multicenter clinical study to evaluate radiographic fusion and clinical outcomes of FIBERGRAFT™ Aeridyan Matrix bone graft substitute in subjects who undergo a 1-3 level instrumented lumbar posterolateral fusion surgery. This clinical study will be conducted at up to 10 clinical sites within the United States.

DETAILED DESCRIPTION:
To evaluate radiographic and clinical outcomes of subjects undergoing a 1-3 level instrumented posterior fusion with DePuy Synthes FIBERGRAFT Aeridyan Matrix or Demineralized Bone Matrix in the posterolateral lumbar spine.

ELIGIBILITY:
INCLUSION CRITERIA

1. Subjects who require a 1-3 level instrumented PLF fusion in the lumbar spine in conjunction with a 1 to 2 consecutive level posterior lumbar interbody fusion procedure between L1-S1.
2. Skeletally mature subjects at least 18 years of age at the time of consenting.
3. Willing to provide voluntary written informed consent prior to participation in the clinical study.

EXCLUSION CRITERIA

1. Subjects who had previous fusion surgery at the index level(s).
2. Requiring a Posterolateral Fusion in the lumbar spine at more than three levels and/or an interbody fusion at more than two levels
3. Subjects who have demonstrated allergy or foreign body sensitivity to the implant or graft material.
4. Pregnant subjects or planning to become pregnant within the next 24 months.
5. Subjects diagnosed with severe osteoporosis which may prevent adequate fixation and thus preclude the use of these or any other orthopedic implant.
6. Subjects diagnosed with severe instabilities, vertebral fractures, spinal tumors.
7. Subjects who have an uncontrolled systemic or metabolic disease which, in the Investigator's opinion, would compromise their health, safety, or ability to participate or follow-up in this clinical study.
8. Subjects requiring use of an implantable bone graft stimulator or external bone graft stimulator.
9. Subjects that have infection or osteomyelitis at the graft site. Any medical or surgical condition that precludes the potential benefit of spinal surgery, in the opinion of the Investigator.
10. Any medical or surgical condition that precludes the potential benefit of spinal surgery, in the opinion of the Investigator.
11. Dependency on pharmaceutical drugs, drug abuse, or alcoholism resulting in a lack of subject cooperation.
12. Subjects unable to comply, and/or in the Investigator's opinion unable to comply, with the requirements of participation in the clinical study.
13. Enhanced Demineralized Bone Matrix product for the grafting control used within the posterolateral spine
14. Use of Bone Morphogenetic Protein (BMP) grafting material within the interbody cage(s).
15. Body Mass Index (BMI) ≥ 45
16. Unilateral posterior instrumentation
17. Subject is currently involved in a workers' compensation claim.
18. Subject has participated in an interventional clinical trial within the last 6 months or plans to participate in an interventional clinical trial within the next 24 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 12 Months
  FIBERGRAFT Aeridyan Matrix percent levels fused at 12 months compared to the grafting control in the posterolateral lumbar spine

SECONDARY OUTCOMES:
Secondary Outcome | 12 Months
  FIBERGRAFT Aeridyan Matrix clinical outcomes (NRS, ODI) change in baseline to 12 months compared to grafting control
Secondary Outcome | 24 months
  FIBERGRAFT Aeridyan Matrix clinical outcomes (NRS, ODI) change in baseline to 24 months compared to grafting control
Secondary Outcome | 6 months
  FIBERGRAFT Aeridyan Matrix percent levels fused at 6 months compared to the grafting control in the posterolateral lumbar spine
Secondary Outcome | 6 months and 12 months
  FIBERGRAFT Aeridyan Matrix percent subjects fused at 6 and at 12 months compared to the grafting control in the posterolateral lumbar spine
Secondary Outcome | Through study completion
  Reoperation/Revision rates of FIBERGRAFT Aeridyan Matrix compared to the grafting control

OTHER OUTCOMES:
Exploratory Endpoint | 6 months
  FIBERGRAFT Aeridyan Matrix percent levels fused at 6 months compared to the grafting control in Cohort B in the posterolateral lumbar spine
Exploratory Endpoint | 12 Months
  FIBERGRAFT Aeridyan Matrix percent levels fused at 12 months compared to the grafting control in Cohort B in the posterolateral lumbar spine
Exploratory Endpoint | 6 months
  FIBERGRAFT Aeridyan Matrix percent subjects fused at 6 months compared to the grafting control in Cohort B in the posterolateral lumbar spine
Exploratory Endpoint | 12 months
  FIBERGRAFT Aeridyan Matrix percent subjects fused at 12 months compared to the grafting control in Cohort B in the posterolateral lumbar spine

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Corrado, Study Chair — DePuy Synthes Products, Inc.
Locations (7):
- United States (7):
  - UC Davis Health System, Sacramento, California
  - University Of Illinois, Chicago, Illinois
  - UK Health Care Kentucky Neuroscience Institute, Lexington, Kentucky
  - Brigham And Women's Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Rothman Orthopaedics Institute, Philadelphia, Pennsylvania
  - UT Health Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No